CLINICAL TRIAL: NCT06798168
Title: Bacteriophage Clinical Trial for Periprosthetic Joint Infection of Multidrug Resistant Pseudomonas Aeruginosa
Status: Available | Type: Expanded Access
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: OLIP1
Record Dates: First submitted 2025-01-21; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Joint Infection
Keywords: Phage therapy; Periprosthetic Joint Infection; Bacteriophage
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: Combining bacteriophage therapy with antibiotics for a case with hip PJI — The treatment plan is to treat the patient with weekly intra-articular injections of a personalized phage therapy cocktail (QDP-PSA-011) for 3 consecutive weeks. This will be associated with antibiotics for 6 weeks.
  Other Names: bacteriophage intra-articular injection

SUMMARY:
This is a single patient study (SPS) that aims to test the bacteriophage treatment as an experimental treatment on a patient suffering from chronic periprosthetic joint infection (PJI) of the right hip. This patients has been suffering from an infection in the right sided hip arthroplasty with a multidrug resistant (MDR) strain of Pseudomonas aeruginosa bacteria. All treatment options for this type of infection have been exhausted. If this patient remains without treatment then there is a high risk of mortality secondary to sepsis and the only remaining surgical option for this patient is a hind quarter amputation which will be a devastating surgery that will largely affect this patients quality of life. However, a large number of published case series have shown the positive impact of combining bacteriophage therapy with antibiotics to achieve a synergistic antibacterial effect and overcome possible resistance development to clear the infection. Therefore we intend to try the bacteriophage therapy on this patients infected hip in the aim to control the infection and improve the patients quality of life.

DETAILED DESCRIPTION:
Total joint replacement (TJR) has revolutionized care provided for patients suffering from disabling joint pain. Unfortunately, periprosthetic joint infection (PJI) remains a devastating complication and the leading cause of failure after TJR. While the current cost in Canada per hip or knee TJR averages $7k CAD, the cost to treat a PJI complication after a hip or knee TJR is five times that amount. In addition, data collected by national and international joint replacement registries demonstrate that the health and economic burden of PJI is a mounting crisis due to the exponential increase in demand for TJR. Current standard treatment for PJI requires multiple surgical revisions of the infected prosthesis in combination with a prolonged course of systemic antibiotic therapy. This standard treatment approach has a failure rate of 20-30%. Unfortunately, this treatment failure is often associated with high rates of psychological distress, limb amputations and death. Debridement Antibiotic and Implant Retention (DAIR) procedure is one of the surgical options that is routinely used to manage PJI, due to its lower risk of morbidity and surgical cost. DAIR is often used for patients who present with an acute PJI or who cannot tolerate a complex implant revision. However, the overall success rate for DAIR is on the lower end of the spectrum, ranging between 60-70%. DAIR failures are often attributed to the residual infection and biofilm burden left behind on the retained implant surface, which cannot be targeted effectively with post-operative systemic antibiotics. Therefore, research has been ongoing to identify non-surgical multidrug resistance (MDR) treatment adjuncts that can synergize the therapeutic effects of antibiotics in PJI care. Numerous preclinical bone and joint infection models have clearly demonstrated such therapeutic benefits using bacteriophages (phages). Phages have the ability to target bacterial cells and breakdown biofilm that it forms on the implant surface. Each bacterial strain tends to have a particular phage that it is susceptible to. Due to this phage specificity and the fact that bacteria can still develop resistance against a single phage, the concept of using a phage cocktail (mixture of 2 or more phage candidates) has been the preferred treatment approach for applying phage therapy. Using a phage cocktail provides a broader spectrum of strain coverage and also makes it harder for the bacteria to develop resistance. Over the past decade, there has been a rise in international interest and effort to translate the antimicrobial therapeutic potential of phages towards this challenging group of patients suffering from bone and joint infections. Published literature has considered phage therapy to be safe for direct administration at the infection site with minimal adverse events provided that the phage preparation administered meets Good Manufacturing Practice (GMP).

In 2023, Suh et al published a comprehensive review summarizing all the PJI clinical cases treated with phage that have been published in English via PubMed from 2010 (1 January) to 2023 (31 March). Only 5 out of 21 patients developed mild adverse events in the form of fevers and transient transaminitis. Considering the heterogeneity of clinical conditions, treatment, and follow-up protocols, 19 out of 21 phage treated cases reported no signs of persistent clinical infection. Ten out of the 19 successful cases were in patients who received a surgical procedure. However, some patients could not go to surgery (2 cases). Both of these phages treated cases reported no adverse events and no signs of persistent clinical infection. A large number of published case series have also recommended combining the use of phage with antibiotics to achieve synergistic antibacterial effect and overcome possible resistance development.

Despite these promising clinical results, there continues to be significant gaps in knowledge which impedes the clinical application of a new treatment paradigm for PJI that incorporates phage therapy. Some of these knowledge gaps revolve around patient selection, phage formulation, treatment protocols, delivery methods and monitoring outcomes. As proposed by Ferry et al., one of the important steps to overcome barriers for the clinical implementation of phage therapy is designing clinical trials with more focused clinical indications to minimize patient heterogeneity and clinical variability.

Despite the abundance of renowned Canadian expertise in phage biology, Canada is significantly lagging in the arena of phage clinical trials. We are aiming to assess the feasibility of a phage therapy clinical trial by going through the single patient study for our patient that has exhausted all the possible avenues of surgical and medical treatment. The next available surgical option for this patient is a hindquarter amputation which will be a devastating surgery for this patient to undergo and provides no quality-of-life prospects at this patient's age. Also, living with active MDR P. aeruginosa without treatment puts the patient at high risk for mortality secondary to sepsis. After reviewing the literature, for such serious infections that have tried all treatment options and have failed to control that infection, the antibacterial resistance leadership group (ARLG)taskforce has determined that phage therapy is generally safe to administer with adverse events rarely reported.

ELIGIBILITY:
Inclusion Criteria:

* Patient is clinically stable and independently mobile
* Patient has been diagnosed with a multidrug resistant chronic bacterial PJI and has exhausted all other non-debilitating treatment options (including DAIR and antibiotic therapy)

Exclusion Criteria:

* Patient has cultured multiple bacteria and it is difficult for physicians to determine which bacteria is causing the disease
* Patient develops a life threatening condition or a condition that leads to deterioration of the patients medical condition and that is unrelated to the known PJI as cerebrovascular accident, angina, cancer.
* Patient's clinical condition is no longer stable and deteriorating for example, if the patient develops sepsis secondary to PJI prior to the commencement of the phage therapy.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- The Ottawa Hospital, Ottawa, Canada

REFERENCES:
- [Background] Suh GA, Ferry T, Abdel MP. Phage Therapy as a Novel Therapeutic for the Treatment of Bone and Joint Infections. Clin Infect Dis. 2023 Nov 2;77(Suppl 5):S407-S415. doi: 10.1093/cid/ciad533. PMID 37932115
- [Background] Ferry T, Kolenda C, Briot T, Souche A, Lustig S, Josse J, Batailler C, Pirot F, Medina M, Leboucher G, Laurent F, On Behalf Of The Lyon Bji Study Group, On Behalf Of The PHAGEinLYON Study Group. Past and Future of Phage Therapy and Phage-Derived Proteins in Patients with Bone and Joint Infection. Viruses. 2021 Dec 2;13(12):2414. doi: 10.3390/v13122414. PMID 34960683
- [Background] Gibb BP, Hadjiargyrou M. Bacteriophage therapy for bone and joint infections. Bone Joint J. 2021 Feb;103-B(2):234-244. doi: 10.1302/0301-620X.103B2.BJJ-2020-0452.R2. PMID 33517726
- [Background] Liu D, Van Belleghem JD, de Vries CR, Burgener E, Chen Q, Manasherob R, Aronson JR, Amanatullah DF, Tamma PD, Suh GA. The Safety and Toxicity of Phage Therapy: A Review of Animal and Clinical Studies. Viruses. 2021 Jun 29;13(7):1268. doi: 10.3390/v13071268. PMID 34209836
- [Background] Hibstu Z, Belew H, Akelew Y, Mengist HM. Phage Therapy: A Different Approach to Fight Bacterial Infections. Biologics. 2022 Oct 6;16:173-186. doi: 10.2147/BTT.S381237. eCollection 2022. PMID 36225325
- [Background] Akanda ZZ, Taha M, Abdelbary H. Current review-The rise of bacteriophage as a unique therapeutic platform in treating peri-prosthetic joint infections. J Orthop Res. 2018 Apr;36(4):1051-1060. doi: 10.1002/jor.23755. Epub 2017 Nov 22. PMID 28971508
- [Background] Suh GA, Lodise TP, Tamma PD, Knisely JM, Alexander J, Aslam S, Barton KD, Bizzell E, Totten KMC, Campbell JL, Chan BK, Cunningham SA, Goodman KE, Greenwood-Quaintance KE, Harris AD, Hesse S, Maresso A, Nussenblatt V, Pride D, Rybak MJ, Sund Z, van Duin D, Van Tyne D, Patel R; Antibacterial Resistance Leadership Group. Considerations for the Use of Phage Therapy in Clinical Practice. Antimicrob Agents Chemother. 2022 Mar 15;66(3):e0207121. doi: 10.1128/AAC.02071-21. Epub 2022 Jan 18. PMID 35041506
- [Background] Scheper H, Gerritsen LM, Pijls BG, Van Asten SA, Visser LG, De Boer MGJ. Outcome of Debridement, Antibiotics, and Implant Retention for Staphylococcal Hip and Knee Prosthetic Joint Infections, Focused on Rifampicin Use: A Systematic Review and Meta-Analysis. Open Forum Infect Dis. 2021 Jul 1;8(7):ofab298. doi: 10.1093/ofid/ofab298. eCollection 2021 Jul. PMID 34258321
- [Background] Bourget-Murray J, Tubin N, Bureau A, Morris J, Ann Azad M, Abdelbary H, Grammatopoulos G, Garceau S. Lower Rates of Reoperation Following Partial or Complete Revision Arthroplasty Compared to Debridement, Antibiotics, and Implant Retention for Early Postoperative and Acute Hematogenous Periprosthetic Hip Infection. J Arthroplasty. 2024 Sep;39(9):2346-2351. doi: 10.1016/j.arth.2024.03.054. Epub 2024 Mar 24. PMID 38531489
- [Background] Taha M, Arnaud T, Lightly TJ, Peters D, Wang L, Chen W, Cook BWM, Theriault SS, Abdelbary H. Combining bacteriophage and vancomycin is efficacious against MRSA biofilm-like aggregates formed in synovial fluid. Front Med (Lausanne). 2023 Jun 9;10:1134912. doi: 10.3389/fmed.2023.1134912. eCollection 2023. PMID 37359001
- [Background] Morcos MW, Kooner P, Marsh J, Howard J, Lanting B, Vasarhelyi E. The economic impact of periprosthetic infection in total knee arthroplasty. Can J Surg. 2021 Mar 5;64(2):E144-E148. doi: 10.1503/cjs.012519. PMID 33666386
- [Background] Akindolire J, Morcos MW, Marsh JD, Howard JL, Lanting BA, Vasarhelyi EM. The economic impact of periprosthetic infection in total hip arthroplasty. Can J Surg. 2020 Jan 29;63(1):E52-E56. doi: 10.1503/cjs.004219. PMID 31995337
- [Background] Matar WY, Jafari SM, Restrepo C, Austin M, Purtill JJ, Parvizi J. Preventing infection in total joint arthroplasty. J Bone Joint Surg Am. 2010 Dec;92 Suppl 2:36-46. doi: 10.2106/JBJS.J.01046. No abstract available. PMID 21123590
- [Background] Kamath AF, Ong KL, Lau E, Chan V, Vail TP, Rubash HE, Berry DJ, Bozic KJ. Quantifying the Burden of Revision Total Joint Arthroplasty for Periprosthetic Infection. J Arthroplasty. 2015 Sep;30(9):1492-7. doi: 10.1016/j.arth.2015.03.035. Epub 2015 Mar 31. PMID 25865815